CLINICAL TRIAL: NCT06522048
Title: SJS/TEN or Other Cutaneous Adverse Eevents Induced by Immune Checkpoint Inhibitors (ICIs) Versus Non-ICIs in Chinese Patients
Brief Title: SJS/TEN or Other Cutaneous Adverse Eevents Induced by Immune Checkpoint Inhibitors (ICIs) vs. Non-ICIs
Status: Completed | Type: Observational
Sponsor: Chao Ji (Other)
Responsible Party: Sponsor-Investigator, Chao Ji, Vice President of the Dermatology Branch of the First Affiliated Hospital of Fujian Medical University, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: Ethical Number [2021]261
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Immune Checkpoint Inhibitor-Induced Dermatitis; Stevens-Johnson Syndrome, Drug-Induced; Toxic Epidermal Necrolysis Due to Drug
MeSH Terms: conditions — Stevens-Johnson Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-immune checkpoint inhibitor (non-ICI) drugs group: Stevens-Johnson Syndrome/Toxic Epidermal Necrolysis (SJS/TEN) induced by non-immune checkpoint inhibitor (non-ICI) drugs
  Interventions: Other: Observational studies do not require intervention
- Immune checkpoint inhibitor (ICIs) group: Stevens-Johnson Syndrome/Toxic Epidermal Necrolysis (SJS/TEN) induced by immune checkpoint inhibitor (ICIs)
  Interventions: Other: Observational studies do not require intervention

INTERVENTIONS:
Other: Observational studies do not require intervention — This is an observational retrospective study and does not require any intervention.

SUMMARY:
Stevens-Johnson Syndrome/Toxic Epidermal Necrolysis (SJS/TEN) is a severe adverse drug reaction, characterized by extensive skin detachment. With the increasing use of immune checkpoint inhibitors (ICIs) in oncology, it is crucial to understand the differences in SJS/TEN induced by ICIs compared to other drugs. This study aims to compare the clinical manifestations and outcomes of Stevens-Johnson Syndrome/Toxic Epidermal Necrolysis (SJS/TEN) or other severity of cutaneous adverse events induced by immune checkpoint inhibitors (ICIs), versus other types of drugs. We analyzed differences in clinical characteristics, treatment methods, outcomes, and survival time and quality of life.

DETAILED DESCRIPTION:
Introduction:

Stevens-Johnson Syndrome/Toxic Epidermal Necrolysis (SJS/TEN) is a severe adverse drug reaction characterized by extensive skin detachment. With the increasing use of immune checkpoint inhibitors (ICIs) in oncology, it is crucial to understand the differences in SJS/TEN induced by ICIs compared to other drugs. This study aims to compare the clinical manifestations and outcomes of Stevens-Johnson Syndrome/Toxic Epidermal Necrolysis (SJS/TEN) or other severity of cutaneous adverse events induced by immune checkpoint inhibitors (ICIs) versus other type drugs. We analyzed differences in clinical characteristics, treatment methods, outcomes, and survival time and quality of life.

Methods:

* Study Design: Retrospective cohort study or cross-sectional study.
* Participants: 60 patients with ICI-induced SJS/TEN and 100 to 500 patients with other drug-induced SJS/TEN.
* Data Collection: Detailed medical records were reviewed to extract information.
* Statistical Analysis: analysis using appropriate statistical tests (e.g., t-test, chi-square test).

Results:

Present the analysis results, highlighting significant differences between the two groups. Use tables and graphs to illustrate key findings.

Conclusion:

We discuss the clinical implications of the findings, potential mechanisms underlying the observed differences, and the relevance to patient management. Summarize the main findings and their significance for clinical practice. Emphasize the need for tailored treatment approaches based on the type of drug causing SJS/TEN.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of SJS/TEN induced by any drugs
* Have the immune-related cutaneous adverse events

Exclusion Criteria:

* Incomplete medical records
* Unknown the specific culprit drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Detailed patient records for SJS/TEN were available in the dermatology inpatient department according to inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2024-05 (Actual); Study Completion 2024-05 (Actual)

PRIMARY OUTCOMES:
Analysis of Clinical Features of Stevens-Johnson Syndrome and Toxic Epidermal Necrolysis Induced by Immune Checkpoint Inhibitors Versus Non-Immune Checkpoint Inhibitors Medications | January 2015 to May 2024
  Present the analysis results, highlighting significant differences between the two groups. Use tables and graphs to illustrate key findings.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerull R, Nelle M, Schaible T. Toxic epidermal necrolysis and Stevens-Johnson syndrome: a review. Crit Care Med. 2011 Jun;39(6):1521-32. doi: 10.1097/CCM.0b013e31821201ed. PMID 21358399
- [Background] Brahmer JR, Lacchetti C, Schneider BJ, Atkins MB, Brassil KJ, Caterino JM, Chau I, Ernstoff MS, Gardner JM, Ginex P, Hallmeyer S, Holter Chakrabarty J, Leighl NB, Mammen JS, McDermott DF, Naing A, Nastoupil LJ, Phillips T, Porter LD, Puzanov I, Reichner CA, Santomasso BD, Seigel C, Spira A, Suarez-Almazor ME, Wang Y, Weber JS, Wolchok JD, Thompson JA; National Comprehensive Cancer Network. Management of Immune-Related Adverse Events in Patients Treated With Immune Checkpoint Inhibitor Therapy: American Society of Clinical Oncology Clinical Practice Guideline. J Clin Oncol. 2018 Jun 10;36(17):1714-1768. doi: 10.1200/JCO.2017.77.6385. Epub 2018 Feb 14. PMID 29442540
- [Background] Zimmermann S, Sekula P, Venhoff M, Motschall E, Knaus J, Schumacher M, Mockenhaupt M. Systemic Immunomodulating Therapies for Stevens-Johnson Syndrome and Toxic Epidermal Necrolysis: A Systematic Review and Meta-analysis. JAMA Dermatol. 2017 Jun 1;153(6):514-522. doi: 10.1001/jamadermatol.2016.5668. PMID 28329382
- [Background] Van Wilpe S, Koornstra R, Den Brok M, De Groot JW, Blank C, De Vries J, Gerritsen W, Mehra N. Lactate dehydrogenase: a marker of diminished antitumor immunity. Oncoimmunology. 2020 Feb 26;9(1):1731942. doi: 10.1080/2162402X.2020.1731942. eCollection 2020. PMID 32158624
- [Background] Lin CC, Chen CB, Wang CW, Hung SI, Chung WH. Stevens-Johnson syndrome and toxic epidermal necrolysis: risk factors, causality assessment and potential prevention strategies. Expert Rev Clin Immunol. 2020 Apr;16(4):373-387. doi: 10.1080/1744666X.2020.1740591. Epub 2020 Apr 2. PMID 32154748